CLINICAL TRIAL: NCT06978595
Title: Primary Colorectal Signet Ring Cell Carcinoma and the Risk of Multiple Primary Gastrointestinal Malignancies: a Retrospective Cohort Based on SEER Database From 2000-2021
Brief Title: Primary Colorectal Signet Ring Cell Carcinoma and the Risk of Multiple Primary Gastrointestinal Malignancies
Status: Completed | Type: Observational
Sponsor: asmaa salama ibrahim (Other)
Responsible Party: Sponsor-Investigator, asmaa salama ibrahim, Resident physician of gastroenterology, Suez Canal University
Organization: Suez Canal University (Other)
Other Study IDs: Z2730
Record Dates: First submitted 2025-04-30; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Carcinoma; Cancer; Signet Ring Adenocarcinoma of the Colon
Keywords: signet ring carcinoma; SEER; Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Carcinoma, Signet Ring Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This original research investigates the critical issue of gastrointestinal (GI) second primary malignancies (SPMs) in patients with signet ring cell carcinoma (SRCC), a rare and aggressive subtype of colorectal cancer. Utilizing the Surveillance, Epidemiology, and End Results (SEER) database, the investigators assessed the risk of GI SPMs, particularly within 2-11 months post-SRCC diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary colorectal SRCC between 2000 and 2021
* Latency exclusion period of two months

Exclusion Criteria:

* patients with unknown age data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with primary colorectal SRCC between 2000 and 2021 were included. Demographic characteristics extracted included race (White, Black, and other races: American Indian/Alaska Native and Asian/Pacific Islander), age (pediatrics: <18 years, young adults: 18-39 years, middle-aged: 40-64 years, elderly: ≥65 years, according to the WHO classification), marital status (married, unmarried, or unknown), and year of diagnosis. Tumor-related variables included stage (in situ, localized, regional, distant, per SEER staging definitions [19]), tumor grade (well-differentiated/grade I, moderately differentiated/grade II, poorly differentiated/grade III, undifferentiated anaplastic/grade IV, and unknown grade), and treatment-related variables (chemotherapy, radiation, and surgery).
Sampling Method: Probability Sample
Enrollment: 8171 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The standardized incidence ratio of developing gastrointestinal second primary malignancies following primary colorectal signet ring cell carcinoma | from Jan, 2000 till Dec, 2021
  The surveillance, epidemiology and End Results (SEER) database was used to calculate the standardized incidence ratio (SIR) as Observed/Expected (O/E) for second primary gastrointestinal malignancies. Patients diagnosed with primary colorectal SRCC between 2000 and 2021 were included. The event was defined as the appearance of an SPM in a different site from the original cancer at a new GI organ (esophagus, stomach, small intestine, cecum, appendix, rectum, anus and anal canal, liver, gallbladder, intrahepatic bile duct, pancreas, retro-peritoneum, and colon).

SECONDARY OUTCOMES:
The excess risk of developing gastrointestinal second primary malignancies following primary colorectal signet ring cell carcinoma | from Jan, 2000 till Dec, 2021
  The excess risk per 10,000 was calculated using SEER*stat software.

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided